CLINICAL TRIAL: NCT03008447
Title: A Randomized, Double-Blind, Placebo-Controlled and Active Comparator, 4 Period Crossover Study to Evaluate the Effect of Lemborexant Versus Placebo and Zolpidem on Postural Stability, Auditory Awakening Threshold, and Cognitive Performance in Healthy Subjects 55 Years and Older
Brief Title: Crossover Study to Evaluate the Effect of Lemborexant Versus Placebo and Zolpidem on Postural Stability, Auditory Awakening Threshold, and Cognitive Performance in Healthy Subjects 55 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: E2006-A001-108
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2017-11

CONDITIONS: Healthy Subjects
Keywords: E2006; postural stability; auditory awakening threshold; cognitive performance; healthy participants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- LEM5; LEM10; PBO; ZOL (Experimental): Participants will receive LEM5 (one lemborexant [LEM] 5 milligram [mg] tablet and one zolpidem [ZOL]-matched placebo [PBO] tablet) in Treatment Period 1. In Treatment Period 2, participants will receive LEM10 (one LEM 10 mg tablet and one ZOL-matched PBO tablet). In Treatment Period 3, participants will receive PBO (one LEM-matched PBO tablet and one ZOL-matched PBO tablet). In Treatment Period 4, participants will receive ZOL (one LEM-matched PBO tablet and one ZOL 6.25 mg tablet).
  Interventions: Drug: LEM5; Drug: LEM10; Drug: ZOL; Drug: PBO
- LEM10; ZOL; LEM5; PBO (Experimental): Participants will receive LEM10, ZOL, LEM5, and PBO in Treatments Periods 1, 2, 3, and 4, respectively.
  Interventions: Drug: LEM5; Drug: LEM10; Drug: ZOL; Drug: PBO
- ZOL; PBO; LEM10; LEM5 (Experimental): Participants will receive ZOL, PBO, LEM10, and LEM5 in Treatment Periods 1, 2, 3, and 4, respectively.
  Interventions: Drug: LEM5; Drug: LEM10; Drug: ZOL; Drug: PBO
- PBO; LEM5; ZOL; LEM10 (Experimental): Participants will receive PBO, LEM5, ZOL, and LEM10 in Treatment Periods 1, 2, 3, and 4, respectively.
  Interventions: Drug: LEM5; Drug: LEM10; Drug: ZOL; Drug: PBO

INTERVENTIONS:
Drug: LEM5 — Single dose of lemborexant 5 mg administered within 5 minutes before bedtime.
Drug: LEM10 — Single dose of lemborexant 10 mg administered within 5 minutes before bedtime.
Drug: ZOL — Single dose of zolpidem 6.25 mg administered within 5 minutes before bedtime.
Drug: PBO — Single dose of placebo administered within 5 minutes before bedtime.

SUMMARY:
E2006-A001-108 is a 4-period crossover study designed to demonstrate that the mean change from baseline in postural stability (worsening) when participants are awakened at approximately 4 hours postdose is significantly less after lemborexant than after zolpidem tartrate extended release following a single-dose administration at bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking female participants, aged 55 years and older, or male participants, aged 65 years and older, at the time of informed consent
* Regular sleep timing and duration, per the following criteria:

  1. Regular time in bed, between 7 and 9 hours as reported at Screening and verified by the Sleep Diary during the Screening Period before the adaptation night such that time in bed is not less than 7 hours or more than 9 hours on more than 2 of the 7 consecutive nights recorded in the Sleep Diary
  2. Regular bedtime, defined as the time the participant attempts to fall asleep, between 22:00 and 01:00 and regular waketime, defined as the time the participant gets out of bed for the day, between 05:00 and 09:00 as reported at Screening and verified by the Sleep Diary during the Screening Period before the adaptation night such that neither bedtime nor waketime is outside of the permitted time windows on more than 2 of the 7 consecutive nights
* Able to detect a 1000 Hertz (Hz) tone at 20 decibels (dB)
* Able to read English at an 8th-grade level

Exclusion Criteria:

* Is a female of childbearing potential Note: All females will be considered to be of childbearing potential unless they are postmenopausal (defined as amenorrheic for at least 12 consecutive months, and are postmenopausal without other known or suspected cause), or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* A current diagnosis of insomnia disorder, sleep-related breathing disorder, periodic limb movements disorder (PLMD), restless legs syndrome, circadian rhythm sleep disorder, narcolepsy, sleep-related violent behavior, sleep-driving, sleep-eating, or symptoms of another parasomnia that in the investigator's opinion make the participant unsuitable for the study
* Has subjective sleep onset latency (sSOL) > 20 minutes or subjective wake after sleep onset (sWASO) > 60 minutes on more than 2 nights as reported on the Sleep Diary during the Screening Period before the adaptation night
* Latency to persistent sleep (LPS) longer than 30 minutes as measured on the PSG on the Baseline night (or repeat Baseline night, if needed)
* Has a sleep onset Rapid eye movement (REM) period, defined as first epoch of stage REM within 15 minutes of sleep onset, as measured on the PSG on either the adaptation night or Baseline night (or repeat Baseline night, if needed)
* Apnea-Hypopnea Index > 15 or Periodic Limb Movement with Arousal Index > 15 as measured on the PSG on the adaptation night
* Comorbid nocturia resulting in frequent need to get out of bed to use the bathroom during the night
* History of fracture due to a fall within the past 5 years
* Evidence of orthostatic hypotension at Screening
* Use of hearing aid or clinically significant hearing loss
* Presence or history of Meniere's disease, labyrinthitis, benign paroxysmal positional vertigo, no recent vertigo from any other cause, no recent dizziness or head injury
* Unable to stand unaided for a minimum of 2 minutes
* At Screening, fails Romberg test in the clinical judgment of the investigator
* Significant vision loss or inability to read computer screen in <80 lumens per square meter (lux) ambient illumination
* History of drug or alcohol dependency or abuse within approximately the previous 2 years or have a positive urine drug screen at Screening or Baseline
* Self-reports consuming more than 14 alcohol-containing drinks per week (females) or 21 alcohol containing drinks per week (males) at Screening
* A prolonged QT/heart rate corrected QT interval (QTc) (QT interval corrected for Fridericia's formula [QTcF] > 450 milliseconds [ms]) as demonstrated by a repeated electrocardiogram (ECG) at Screening (repeated only if initial ECG indicates a QTcF interval > 450 ms)
* Any suicidal ideation at Screening or within 6 months of Screening or any lifetime suicidal behavior
* Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal, psychiatric or neurological disease, malignancy other than basal cell carcinoma, or chronic pain) or condition that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 half lives, whichever is longer, before the Baseline night
* Scheduled for surgery during the study
* Transmeridian travel across more than 3 time zones in the 2 weeks before the first Baseline night, or plans to travel more than 3 time zones during the study.
* Currently enrolled in another clinical trial or used any investigational drug or device within 28 days or 5 half lives, whichever is longer preceding informed consent
* Hypersensitivity to lemborexant or zolpidem or any of their excipients
* Active viral hepatitis (B or C) as demonstrated by positive serology
* Previous exposure to lemborexant or suvorexant

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Change from time-matched baseline in postural stability for LEM5 and LEM10 compared to zolpidem (ZOL) at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
  Magnitude of body sway upon being awakened at approximately 4 hours after receiving lemborexant 5 milligrams (mg) (LEM5), lemborexant 10 mg (LEM10), zolpidem 6.25 mg, or placebo.

SECONDARY OUTCOMES:
Change from time-matched baseline in postural stability for LEM5 and LEM10 compared to ZOL and placebo (PBO) at approximately 8 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline in postural stability for LEM5 and LEM10 compared to PBO at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline in auditory awakening threshold (AAT) for LEM5 and LEM10 compared to ZOL and PBO at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from power of attention for LEM5 and LEM10 compared to ZOL and PBO at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from power of attention for LEM5 and LEM10 compared to ZOL and PBO at approximately 8 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from continuity of attention for LEM5 and LEM10 compared to ZOL and PBO at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from continuity of attention for LEM5 and LEM10 compared to ZOL and PBO at approximately 8 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from quality of memory for LEM5 and LEM10 compared to ZOL and PBO at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from quality of memory for LEM5 and LEM10 compared to ZOL and PBO at approximately 8 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from speed of memory retrieval for LEM5 and LEM10 compared to ZOL and PBO at approximately 4 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Change from time-matched baseline on summary variables from speed of memory retrieval for LEM5 and LEM10 compared to ZOL and PBO at approximately 8 hours postdose | approximately 4 hours postdose at each of 4 single-dose treatment periods (up to 43 days)
Number of participants with any serious adverse event and number of participants with any non-serious adverse event | up to 72 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NeuroTrials Research, Inc, Atlanta, Georgia
  - Clinilabs, Inc, New York, New York
  - Wake Research Assoicates, LLC, Raleigh, North Carolina
  - Community Research Management Associates d/b/a CTI Clinical Research Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Gotfried MH, Auerbach SH, Dang-Vu TT, Mishima K, Kumar D, Moline M, Malhotra M. Efficacy and safety of insomnia treatment with lemborexant in older adults: analyses from three clinical trials. Drugs Aging. 2024 Sep;41(9):741-752. doi: 10.1007/s40266-024-01135-8. Epub 2024 Aug 9. PMID 39120786
- [Derived] Murphy P, Kumar D, Zammit G, Rosenberg R, Moline M. Safety of lemborexant versus placebo and zolpidem: effects on auditory awakening threshold, postural stability, and cognitive performance in healthy older participants in the middle of the night and upon morning awakening. J Clin Sleep Med. 2020 May 15;16(5):765-773. doi: 10.5664/jcsm.8294. Epub 2020 Feb 6. PMID 32022664